CLINICAL TRIAL: NCT00367380
Title: Evaluation of Reproducibility of a Sporozoite Challenge Model for Plasmodium Vivax in Human Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Malaria Vaccine and Drug Development Center (Other)
Collaborators: Fundacion Clinica Valle del Lili (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MVDC-2006-004
Record Dates: First submitted 2006-08-19; First posted 2006-08-22 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2021-02

CONDITIONS: MALARIA; FEVER; Sweating Fever; Chills; ANEMIA
Keywords: Malaria; Sporozoite; Challenge Model; Plasmodium vivax; Human Volunteers
MeSH Terms: conditions — Malaria; Fever; Chills; Anemia; Malaria, Vivax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): 6 volunteers to be challenged with the infected with +/-3 mosquito bites from batch 413ABM
  Interventions: Other: 413ABM
- Group 2 (Experimental): 6 volunteers to be challenged with the infected with +/-3 mosquito bites from batch 414WRR
  Interventions: Other: 414WRR
- Group 3 (Experimental): 6 volunteers to be challenged with the infected with +/-3 mosquito bites from batch 418JAL
  Interventions: Other: 418JAL

INTERVENTIONS:
Other: 413ABM — +/- 3 bites of Anopheles albimanus mosquitoes infected through membrane feeding with blood of the P. vivax infected volunteers 413ABM
  Arms: Group 1
Other: 414WRR — +/- 3 bites of Anopheles albimanus mosquitoes infected through membrane feeding with blood of the P. vivax infected volunteers 414WRR
  Arms: Group 2
Other: 418JAL — +/- 3 bites of Anopheles albimanus mosquitoes infected through membrane feeding with blood of the P. vivax infected volunteers 418JAL
  Arms: Group 3

SUMMARY:
The study is a randomized open label clinical trial to verify the reproducibility of a sporozoite challenge model for Plasmodium vivax in humans. The verification of the reproducibility of such a model will make it possible to evaluate the efficacy of candidate P. vivax vaccines in Phase 2a trials. The study is divided into two successive steps:

Step A Parasite Blood Donation: Volunteers will be recruited passively from a group of patients who present with active P. vivax infection and accept to donate infected blood. Samples of P. vivax infected blood will be collected and will be screened for infectious diseases, according to standard blood bank procedures. Colonized Anopheles albimanus mosquitoes will be fed with this blood using a Membrane Feeding Assay (MFA). Sixteen (16) days after, selected positive mosquito batches will be used for step B.

Step B Challenge: After informed consent signature, a total of 18 healthy volunteers will be randomly allocated to Groups 1, 2 and 3, of 6 volunteers each and will be challenged with the bite of 3±1, P. vivax infected mosquitoes. Each group will be exposed to a different isolated parasite. Volunteers will be closely monitored post infection, and will be treated as soon as blood infection becomes patent as ascertained by microscopic examination of thick blood smears (TBS). Comparison of data obtained in the three different groups will be used to determine reproducibility of challenge model.

Primary objective: To demonstrate that naïve human volunteers can be safely and reproducibly infected by the bite of An. albimanus mosquitoes carrying P. vivax sporozoites in their salivary glands.

Secondary objective: To determine the influence of the type of parasite isolated on reproducibility and safety of the challenge model with P. vivax in human volunteers

Hypothesis:It is possible to safely develop a reproducible P. vivax infection in human volunteers using P. vivax experimentally infected An. albimanus mosquitoes.

DETAILED DESCRIPTION:
Study design

A randomized, open-label clinical trial was designed to standardize a P. vivax sporozoite challenge model in malaria-naïve volunteers, specifically, the relationship between the number of infectious mosquito bites and the likelihood of developing patent parasitemia detectable by Giemsa-stained thick blood smear (TBS). The study was divided into two steps. Step A was designed to produce mature P. vivax sporozoites suitable for inoculation into humans; and Step B was designed to assess the safety and reproducibility of the sporozoite challenge. For Step A, patients with infective P. vivax gametocytes detected by TBS were recruited from the outpatient clinics at the Immunology Institute (IDIV) in Cali and Buenaventura, Colombia. Patients donated 35 mL of whole blood, which was screened for co-infections that could potentially represent a threat to the health of volunteers. The blood was then artificially fed to Anopheles mosquitoes.14 For Step B, malaria-naive subjects were exposed to the bites of 3 ± 1, 6 ± 1, or 9 ± 1 infected mosquitoes to determine the prepatent period of the infection and its reproducibility.

Blood donation and blood quality assurance

The EDTA vacutainer tubes (Becton Dickinson, Franklin Lakes, NJ) were used to collect 35 mL of whole blood from each infected patient, which were divided into two aliquots: a 15 mL sample for mosquito feeding and a 20 mL sample that was transported to the blood bank of the Valle del Lili Clinic for routine screening for a panel of common infectious agents (viral, bacterial, parasitic), including confirmation of Plasmodium species ( P. vivax, P. falciparum, P. malariae) by polymerase chain reaction (PCR) (Table 2).15 The rationale behind the blood screening and direct mosquito feeding on human volunteers was based on two premises: 1) standard blood bank screening is universally accepted as a safety procedure that ensures that no pathogens are transmitted from human-to-human during a blood transfusion. Therefore, blood samples determined to be negative for pathogens other than P. vivax by standard blood bank screening should be safe enough to be transferred from human-to-human through a mosquito bite. 2) Anopheles mosquitoes have not been reported to trans mit any pathogen other than Plasmodium. Before the study, we carried out an extensive bibliographic search and consulted with U.S. and Colombian experts on virology, parasitology, and entomology about potential pathogens that might be transmitted by Anopheles and could represent a threat for the volunteers exposed to challenge. There was a consensus that as yet no other pathogen had been reported to be transmitted by Anopheles mosquitoes, including those comprised in the blood bank screening. However, mosquitoes were discarded using a biosafety procedure if after feeding blood was confirmed to have any co-infection.

Mosquito infection

Anopheles albimanus mosquitoes Buenaventura strain, have been reared under laboratory conditions at IDIV in Cali for about 10 years. This mosquito colony has been successfully used to regularly produce sporozoites14,16 and for studies on malaria transmission-blocking immunity.17 Here, mosquitoes were fed within 2-3 hours after the P. vivax-infected blood (gametocytemia ≥ 0.1%) was collected in Buenaventura. The 15 mL blood was centrifuged at 500 × g for 5 minutes at room temperature, plasma was removed, and cells were washed once with RPMI 1640 medium (Gibco Cell Culture Systems, Invitrogen, Grand Island, NY ). Parasitized erythrocytes were reconstituted to 50% hematocrit with pooled human AB non-immune, complement-inactivated serum obtained from the Red Cross blood bank and were used to infect lots of 4,000 female mosquitoes (3-4 days old) using a water-jacketed membrane apparatus at 37°C, described previously.14 Infected mosquitoes were maintained under strict biosafety conditions at 27 ± 1°C and relative humidity of 82% and a sugar solution supplemented with 0.05% para-aminobenzoic-acid was provided.18 Samples of fed mosquitoes were dissected and microscopically examined 7-8 days after the blood meal to determine the presence of oocysts in the midgut, and on Days 14 and 15 to assess the presence of sporozoites in salivary glands.19 Mosquito infections were graded as 1+ (1-10 spz), 2+ (11-100 spz), 3+ (101-1000 spz), and 4+ (> 1001 spz).7

Sporozoite challenge

The proposed infective biting dose was to be 3, 6, and 9 mosquitoes, respectively. However, a range of plus or minus one bite per dose was allowed. Therefore, screen-meshed boxes (7 × 7 × 7 cm) were filled with 4, 7, and 10 mosquitoes, to have a better chance of achieving the targeted mosquito dose in a single biting round. Participants who did not complete the minimal targeted dose were subjected to a second round of biting. Eighteen malaria-naïve volunteers were randomly assigned to one of three groups (N = 6) and were exposed by group, from the fewest (3 bites) to the greatest (9 bites) number of bites. Sporozoite challenge was carried out under strict adherence to experimental protocol in a secure room in the entomology unit at the IDIV. Volunteers were asked not to use any topical chemicals (e.g., soap, deodorant, perfume) that could affect mosquito feeding. Mosquitoes were allowed to bite the flexor side of the forearm for a 10 to 15-minute period, previously determined to be sufficient for full An. albimanus engorgement. After biting, all mosquitoes were dissected to confirm the presence of blood meal and sporozoites. Mosquitoes were considered positive if any number of sporozoites (> 1) was detected microscopically. Study participants were observed for 1 hour at the entomology unit, followed up by phone 8 hours later, and examined again 24 hours thereafter to assess the response to challenge.

Malaria diagnosis and patient follow-up

From Day 7 post-challenge onward, volunteers had daily follow-up visits during which symptoms and signs of malaria were assessed and blood was collected for TBS and Plasmodium PCR (the latter performed retrospectively).

The TBS were performed using 50 μL of whole blood collected by finger prick that were spread over a rectangular area of approximately 1.5 sq cm and were stained with freshly prepared 10% Giemsa stain.20 A total of 300 microscopic fields were examined before a slide was considered negative. When TBS were found positive, parasitemia was quantified by estimating the number of parasites counted in presence of 300 leukocytes and calculating absolute parasitemia according the leukocyte counts per μL. Smears were read by experienced microscopists and a random sample of TBS was subjected to quality control by a microscopist from the malaria control program.

Participants were treated with anti-malarial drugs as soon as parasites were detected by TBS. Treatment consisted of chloroquine (1,500 mg chloroquine base provided orally in divided doses: 600 mg initially followed by 450 mg given 24 and 48 hours later) and primaquine (two 15 mg doses given once per day for 14 days). Volunteers were provided with intravenous fluids, analgesics, and antiemetics as needed. Signs and symptoms consistent with malaria were assessed by clinical examination and were graded 1-5 according to their severity following the National Cancer Institute (NCI) criteria for adverse events (CTCAE ) as follows: Grade 1 = Low, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Serious, and Grade 5 = Death. Pruritus was graded from 1 to 3 (1 = mild or localized; 2 = intense or widespread; and 3 = intense or widespread and interfering with activities of daily living). Because there is no common terminology AE agreement, for edema and erythema following mosquito bites, an adaptation from the CTCAE v 3 for "injection site/extravasation changes" was used as follows: Grade 1 = local pain/edema and erythema; Grade 2 = pain or swelling with inflammation or phlebitis; Grade 3 = ulceration or necrosis. Pain was scored as Grade 1 = mild not interfering with function; Grade 2 = moderate pain (pain or analgesics interfering with function, but not interfering with activities of daily living); Grade 3 = severe pain (pain or analgesics severely interfering with activities of daily living).

Clinical laboratory tests

Clinical laboratory screening in -clouding an electrocardiogram confirmed the health status of volunteers 1 month before challenge and after the study was completed (Table 1). Any abnormality found in the electrocardiogram was considered as an exclusion criterion. Tests for hemoglobin, white blood cell count, platelet count, and total bilirubin were performed again on Days 11 and 53 post-challenge.

Statistical methods

Sample size (N = 6 per group) was based on the minimum number of individuals that would be allowed to observe the occurrence of rarer events (e.g., events that occur in approximately 5% of individuals) with reasonable probability based on a binomial assumption. The overall sample size of 18 would be sufficient to detect even rare events. A titration of mosquito bites (biting doses) was established; beginning with that arbitrarily considered the minimum number required causing an infection. Prepatent periods and duration of symptoms were expressed as geometric means. Differences among the groups were estimated by the Kruskal-Wallis test, and were considered statistically significant at P values less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult male or non-pregnant females (18-45 years of age).
* Capacity to sign a free informed consent form of participation along with two witnesses.
* Use of adequate contraceptive method from the initiation of the study until three months after sporozoite challenge.
* No plans to travel to malaria endemic areas during the course of the study (a year).
* No plans to travel outside the study area from the 7th day until 31st day after the challenge.
* Reachable by phone during the whole study period.
* Able to participate during the whole study period.

Exclusion Criteria:

* Are less than 18 and over 45 years of age.
* Are female who is pregnant at serum positive B-HCG screening, planning to become pregnant or who is nursing.
* Have a Duffy negative phenotype.
* Have a G-6-PD deficiency or any other hemoglobinopathy.
* Current or past infection with any species of malaria as demonstrated by a positive TBS on screening or history of a documented positive blood smear. P. vivax IFAT of 1
* Have a known history of allergy to antimalarial drugs or immediate type hypersensitivity reactions to mosquito bites.
* Clinical or laboratory evidence of significant systemic disease, including hepatic, renal, cardiac, immunologic or hematological disease, HIV positive or have any other known immunodeficiency (including receiving immunosuppressive therapy or a history of splenectomy); infected with hepatitis B or C virus; have a history of autoimmune disease (including inflammatory bowel disease, hemolytic anemia, autoimmune hepatitis, rheumatoid arthritis, lupus, etc.) or connective tissue disease or have any other serious underlying medical condition.
* Clinically significant laboratory abnormalities as determined by the Investigator(s).
* Plan to have surgery between enrollment and the end of the challenge follow-up.
* Previous history of alcoholism or drugs use which interfere with social activities of the volunteer
* Have any other conditions that are determined by at least two concurring investigators that may interfere with the capacity to provide free and willing informed consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2006-12; Primary Completion 2006-12 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Socrates Herrera, MD, Principal Investigator — Director
Locations (1):
- Malaria Vaccine and Drug Development Center, Cali, Valle del Cauca Department, Colombia

REFERENCES:
- [Background] Arevalo-Herrera M, Roggero MA, Gonzalez JM, Vergara J, Corradin G, Lopez JA, Herrera S. Mapping and comparison of the B-cell epitopes recognized on the Plasmodium vivax circumsporozoite protein by immune Colombians and immunized Aotus monkeys. Ann Trop Med Parasitol. 1998 Jul;92(5):539-51. PMID 9797827
- [Background] Arevalo-Herrera M, Herrera S. Plasmodium vivax malaria vaccine development. Mol Immunol. 2001 Dec;38(6):443-55. doi: 10.1016/s0161-5890(01)00080-3. PMID 11741694
- [Background] Arevalo-Herrera M, Castellanos A, Yazdani SS, Shakri AR, Chitnis CE, Dominik R, Herrera S. Immunogenicity and protective efficacy of recombinant vaccine based on the receptor-binding domain of the Plasmodium vivax Duffy binding protein in Aotus monkeys. Am J Trop Med Hyg. 2005 Nov;73(5 Suppl):25-31. doi: 10.4269/ajtmh.2005.73.5_suppl.0730025. PMID 16291763
- [Background] Arevalo-Herrera M, Solarte Y, Zamora F, Mendez F, Yasnot MF, Rocha L, Long C, Miller LH, Herrera S. Plasmodium vivax: transmission-blocking immunity in a malaria-endemic area of Colombia. Am J Trop Med Hyg. 2005 Nov;73(5 Suppl):38-43. doi: 10.4269/ajtmh.2005.73.5_suppl.0730038. PMID 16291765
- [Background] Arevalo-Herrera M, Solarte Y, Yasnot MF, Castellanos A, Rincon A, Saul A, Mu J, Long C, Miller L, Herrera S. Induction of transmission-blocking immunity in Aotus monkeys by vaccination with a Plasmodium vivax clinical grade PVS25 recombinant protein. Am J Trop Med Hyg. 2005 Nov;73(5 Suppl):32-7. doi: 10.4269/ajtmh.2005.73.32. PMID 16291764
- [Background] Baird JK, Tiwari T, Martin GJ, Tamminga CL, Prout TM, Tjaden J, Bravet PP, Rawlins S, Ferrel M, Carucci D, Hoffman SL. Chloroquine for the treatment of uncomplicated malaria in Guyana. Ann Trop Med Parasitol. 2002 Jun;96(4):339-48. doi: 10.1179/000349802125001023. PMID 12171615
- [Background] Ballou WR, Arevalo-Herrera M, Carucci D, Richie TL, Corradin G, Diggs C, Druilhe P, Giersing BK, Saul A, Heppner DG, Kester KE, Lanar DE, Lyon J, Hill AV, Pan W, Cohen JD. Update on the clinical development of candidate malaria vaccines. Am J Trop Med Hyg. 2004 Aug;71(2 Suppl):239-47. PMID 15331843
- [Background] Baton LA, Ranford-Cartwright LC. How do malaria ookinetes cross the mosquito midgut wall? Trends Parasitol. 2005 Jan;21(1):22-8. doi: 10.1016/j.pt.2004.11.001. PMID 15639737
- [Background] Blair S, Lopez ML, Pineros JG, Alvarez T, Tobon A, Carmona J. [Therapeutic efficacy of 3 treatment protocols for non-complicated Plasmodium falciparum malaria, Antioquia, Colombia, 2002]. Biomedica. 2003 Sep;23(3):318-27. Spanish. PMID 14582335
- [Background] Blow JA, Turell MJ, Walker ED, Silverman AL. Post-bloodmeal diuretic shedding of hepatitis B virus by mosquitoes (Diptera: Culicidae). J Med Entomol. 2002 Jul;39(4):605-12. doi: 10.1603/0022-2585-39.4.605. PMID 12144291
- [Background] 11. Bosman, A., Delacollette, C., Olumese, P., Ridley, RG., Rietveld, R., Shretta, R.,Teklehaimanot, A. The use of antimalarial drugs. Report of an Informal Consultation. Roll Back Malaria. WHO. 2001.
- [Background] Chauhan VS, Bhardwaj D. Current status of malaria vaccine development. Adv Biochem Eng Biotechnol. 2003;84:143-82. doi: 10.1007/3-540-36488-9_5. PMID 12934936
- [Background] Chappel JA, Rogers WO, Hoffman SL, Kang AS. Molecular dissection of the human antibody response to the structural repeat epitope of Plasmodium falciparum sporozoite from a protected donor. Malar J. 2004 Jul 29;3:28. doi: 10.1186/1475-2875-3-28. PMID 15283866
- [Background] Chotivanich K, Silamut K, Udomsangpetch R, Stepniewska KA, Pukrittayakamee S, Looareesuwan S, White NJ. Ex-vivo short-term culture and developmental assessment of Plasmodium vivax. Trans R Soc Trop Med Hyg. 2001 Nov-Dec;95(6):677-80. doi: 10.1016/s0035-9203(01)90113-0. PMID 11816444
- [Background] Chulay JD, Schneider I, Cosgriff TM, Hoffman SL, Ballou WR, Quakyi IA, Carter R, Trosper JH, Hockmeyer WT. Malaria transmitted to humans by mosquitoes infected from cultured Plasmodium falciparum. Am J Trop Med Hyg. 1986 Jan;35(1):66-8. doi: 10.4269/ajtmh.1986.35.66. PMID 3511753
- [Background] Church LW, Le TP, Bryan JP, Gordon DM, Edelman R, Fries L, Davis JR, Herrington DA, Clyde DF, Shmuklarsky MJ, Schneider I, McGovern TW, Chulay JD, Ballou WR, Hoffman SL. Clinical manifestations of Plasmodium falciparum malaria experimentally induced by mosquito challenge. J Infect Dis. 1997 Apr;175(4):915-20. doi: 10.1086/513990. PMID 9086149
- [Background] Clyde DF, McCarthy VC, Miller RM, Hornick RB. Specificity of protection of man immunized against sporozoite-induced falciparum malaria. Am J Med Sci. 1973 Dec;266(6):398-403. doi: 10.1097/00000441-197312000-00001. No abstract available. PMID 4590095
- [Background] Clyde DF. Immunization of man against falciparum and vivax malaria by use of attenuated sporozoites. Am J Trop Med Hyg. 1975 May;24(3):397-401. doi: 10.4269/ajtmh.1975.24.397. PMID 808142
- [Background] Clyde DF. Immunity to falciparum and vivax malaria induced by irradiated sporozoites: a review of the University of Maryland studies, 1971-75. Bull World Health Organ. 1990;68 Suppl(Suppl):9-12. PMID 2094597
- [Background] Cogswell FB. The hypnozoite and relapse in primate malaria. Clin Microbiol Rev. 1992 Jan;5(1):26-35. doi: 10.1128/CMR.5.1.26. PMID 1735093
- [Background] Collins WE, Jeffery GM. Primaquine resistance in Plasmodium vivax. Am J Trop Med Hyg. 1996 Sep;55(3):243-9. doi: 10.4269/ajtmh.1996.55.243. PMID 8842108
- [Background] Danis M. [Therapeutic advances against malaria in 2003]. Med Trop (Mars). 2003;63(3):267-70. French. PMID 14579464
- [Background] Doolan DL, Hoffman SL. Nucleic acid vaccines against malaria. Chem Immunol. 2002;80:308-21. doi: 10.1159/000058851. No abstract available. PMID 12058647
- [Background] Duarte EC, Pang LW, Ribeiro LC, Fontes CJ. Association of subtherapeutic dosages of a standard drug regimen with failures in preventing relapses of vivax malaria. Am J Trop Med Hyg. 2001 Nov;65(5):471-6. doi: 10.4269/ajtmh.2001.65.471. PMID 11716100
- [Background] Edelman R, Hoffman SL, Davis JR, Beier M, Sztein MB, Losonsky G, Herrington DA, Eddy HA, Hollingdale MR, Gordon DM, et al. Long-term persistence of sterile immunity in a volunteer immunized with X-irradiated Plasmodium falciparum sporozoites. J Infect Dis. 1993 Oct;168(4):1066-70. doi: 10.1093/infdis/168.4.1066. PMID 8376823
- [Background] Egan JE, Hoffman SL, Haynes JD, Sadoff JC, Schneider I, Grau GE, Hollingdale MR, Ballou WR, Gordon DM. Humoral immune responses in volunteers immunized with irradiated Plasmodium falciparum sporozoites. Am J Trop Med Hyg. 1993 Aug;49(2):166-73. doi: 10.4269/ajtmh.1993.49.166. PMID 8357078
- [Background] FAIRLEY NH. Sidelights on malaria in man obtained by subinoculation experiments. Trans R Soc Trop Med Hyg. 1947 May;40(5):621-76. doi: 10.1016/0035-9203(47)90025-4. No abstract available. PMID 20243883
- [Background] Fernández, O.,Manzano, M.R, Murrain, B., Blanco P., Zamora F., Jordan, A. Palacios, R., Velez, D., Arevalo-Herrera, M., Herrera, S. Development of a sporozoite challenge model for Plasmodium vivax in human volunteers. ASTMH. Annual Metting 54th. 2005.
- [Background] Fryauff DJ, Baird JK, Basri H, Sumawinata I, Purnomo, Richie TL, Ohrt CK, Mouzin E, Church CJ, Richards AL, et al. Randomised placebo-controlled trial of primaquine for prophylaxis of falciparum and vivax malaria. Lancet. 1995 Nov 4;346(8984):1190-3. doi: 10.1016/s0140-6736(95)92898-7. PMID 7475658
- [Background] Genton B, Corradin G. Malaria vaccines: from the laboratory to the field. Curr Drug Targets Immune Endocr Metabol Disord. 2002 Oct;2(3):255-67. doi: 10.2174/1568008023340613. PMID 12476490
- [Background] George FW 4th, Law JL, Rich KA, Martin WJ. Identification of a T-cell epitope on the circumsporozoite protein of Plasmodium vivax. Infect Immun. 1990 Feb;58(2):575-8. doi: 10.1128/iai.58.2.575-578.1990. PMID 1688828
- [Background] Glynn JR. Infecting dose and severity of malaria: a literature review of induced malaria. J Trop Med Hyg. 1994 Oct;97(5):300-16. PMID 7932927
- [Background] Glynn JR, Bradley DJ. Inoculum size, incubation period and severity of malaria. Analysis of data from malaria therapy records. Parasitology. 1995 Jan;110 ( Pt 1):7-19. doi: 10.1017/s0031182000080999. PMID 7845714
- [Background] Glynn JR, Collins WE, Jeffery GM, Bradley DJ. Infecting dose and severity of falciparum malaria. Trans R Soc Trop Med Hyg. 1995 May-Jun;89(3):281-3. doi: 10.1016/0035-9203(95)90540-5. PMID 7660433
- [Background] Golenda CF, Li J, Rosenberg R. Continuous in vitro propagation of the malaria parasite Plasmodium vivax. Proc Natl Acad Sci U S A. 1997 Jun 24;94(13):6786-91. doi: 10.1073/pnas.94.13.6786. PMID 9192643
- [Background] Good MF, Pombo D, Quakyi IA, Riley EM, Houghten RA, Menon A, Alling DW, Berzofsky JA, Miller LH. Human T-cell recognition of the circumsporozoite protein of Plasmodium falciparum: immunodominant T-cell domains map to the polymorphic regions of the molecule. Proc Natl Acad Sci U S A. 1988 Feb;85(4):1199-203. doi: 10.1073/pnas.85.4.1199. PMID 2448793
- [Background] Grassi, B., Bignami, A., Bastianelli, G. Ulteriori ricerche sul ciclo dei parassiti malarici umani nel corpo del zanzarone. Atti Reale Accademia dei Lincei. 1899.5:8-21.
- [Background] Hermsen CC, de Vlas SJ, van Gemert GJ, Telgt DS, Verhage DF, Sauerwein RW. Testing vaccines in human experimental malaria: statistical analysis of parasitemia measured by a quantitative real-time polymerase chain reaction. Am J Trop Med Hyg. 2004 Aug;71(2):196-201. PMID 15306710
- [Background] Safety and immunogenecity of a Plasmodium vivax circumsporozoite protein-derived synthetic vaccine in two Montanide ISA formulations.2006a. Manuscrito en preparacion.
- [Background] Herrera S, Bonelo A, Perlaza BL, Fernandez OL, Victoria L, Lenis AM, Soto L, Hurtado H, Acuna LM, Velez JD, Palacios R, Chen-Mok M, Corradin G, Arevalo-Herrera M. Safety and elicitation of humoral and cellular responses in colombian malaria-naive volunteers by a Plasmodium vivax circumsporozoite protein-derived synthetic vaccine. Am J Trop Med Hyg. 2005 Nov;73(5 Suppl):3-9. doi: 10.4269/ajtmh.2005.73.3. PMID 16291760
- [Background] Herrera MA, de Plata C, Gonzalez JM, Corradin G, Herrera S. Immunogenicity of multiple antigen peptides containing Plasmodium vivax CS epitopes in BALB/c mice. Mem Inst Oswaldo Cruz. 1994;89 Suppl 2:71-6. doi: 10.1590/s0074-02761994000600017. PMID 7565136
- [Background] Herrera S, De Plata C, Gonzalez M, Perlaza BL, Bettens F, Corradin G, Arevalo-Herrera M. Antigenicity and immunogenicity of multiple antigen peptides (MAP) containing P. vivax CS epitopes in Aotus monkeys. Parasite Immunol. 1997 Apr;19(4):161-70. doi: 10.1046/j.1365-3024.1997.d01-193.x. PMID 9149283
- [Background] Herrera S, Escobar P, de Plata C, Avila GI, Corradin G, Herrera MA. Human recognition of T cell epitopes on the Plasmodium vivax circumsporozoite protein. J Immunol. 1992 Jun 15;148(12):3986-90. PMID 1376347
- [Background] Herrera, S., Manzano, M., Fernandez, O., Solarte, Y., Rocha, L., Vergara, J., Bermans, M., Acuña, L., Londoño, C., Palacios, R., Rincon, A., Yansot, MF., Arevalo-Herrera, M. Establishment of a sporozoite challenge model for Plasmodium vivax in human volunteers. 2006b. Manuscrito en preparación.
- [Background] Herrera S, Perlaza BL, Bonelo A, Arevalo-Herrera M. Aotus monkeys: their great value for anti-malaria vaccines and drug testing. Int J Parasitol. 2002 Dec 4;32(13):1625-35. doi: 10.1016/s0020-7519(02)00191-1. PMID 12435447
- [Background] Herrington D, Davis J, Nardin E, Beier M, Cortese J, Eddy H, Losonsky G, Hollingdale M, Sztein M, Levine M, et al. Successful immunization of humans with irradiated malaria sporozoites: humoral and cellular responses of the protected individuals. Am J Trop Med Hyg. 1991 Nov;45(5):539-47. doi: 10.4269/ajtmh.1991.45.539. PMID 1951863
- [Background] Hisaeda H, Yasutomo K. Development of malaria vaccines that block transmission of parasites by mosquito vectors. J Med Invest. 2002 Aug;49(3-4):118-23. PMID 12323000
- [Background] Hoffman SL. Experimental challenge of volunteers with malaria. Ann Intern Med. 1997 Aug 1;127(3):233-5. doi: 10.7326/0003-4819-127-3-199708010-00010. No abstract available. PMID 9245231
- [Background] Hoffman SL, Goh LM, Luke TC, Schneider I, Le TP, Doolan DL, Sacci J, de la Vega P, Dowler M, Paul C, Gordon DM, Stoute JA, Church LW, Sedegah M, Heppner DG, Ballou WR, Richie TL. Protection of humans against malaria by immunization with radiation-attenuated Plasmodium falciparum sporozoites. J Infect Dis. 2002 Apr 15;185(8):1155-64. doi: 10.1086/339409. Epub 2002 Apr 1. PMID 11930326
- [Background] Hurtado S, Salas ML, Romero JF, Zapata JC, Ortiz H, Arevalo-Herrera M, Herrera S. Regular production of infective sporozoites of Plasmodium falciparum and P. vivax in laboratory-bred Anopheles albimanus. Ann Trop Med Parasitol. 1997 Jan;91(1):49-60. doi: 10.1080/00034983.1997.11813111. PMID 9093429
- [Background] Jordan, A., Cellular and humoral response of P vivax irradiated sporozoites in Aotus monkeys. Am. J. Trop. Med Hyg., 2006 .Manuscrito en preparación.
- [Background] Krotoski WA. The hypnozoite and malarial relapse. Prog Clin Parasitol. 1989;1:1-19. PMID 2491691
- [Background] Luke TC, Hoffman SL. Rationale and plans for developing a non-replicating, metabolically active, radiation-attenuated Plasmodium falciparum sporozoite vaccine. J Exp Biol. 2003 Nov;206(Pt 21):3803-8. doi: 10.1242/jeb.00644. PMID 14506215
- [Background] Manzano, M.R, Rocha, L., Hurtado, Solarte, Y., Arévalo-Herrera, M., Herrera, S., Development of a sporozoite challenge model of naïve voluntieers using Anopheles albimanus infected with Plasmodium vivax. 2006. Manuscrito en preparación.
- [Background] McCarthy VC, Clyde DF. Plasmodium vivax: correlation of circumsporozoite precipitation (CSP) reaction with sporozoite-induced protective immunity in man. Exp Parasitol. 1977 Feb;41(1):167-71. doi: 10.1016/0014-4894(77)90142-4. No abstract available. PMID 320027
- [Background] McGready R, Thwai KL, Cho T, Samuel, Looareesuwan S, White NJ, Nosten F. The effects of quinine and chloroquine antimalarial treatments in the first trimester of pregnancy. Trans R Soc Trop Med Hyg. 2002 Mar-Apr;96(2):180-4. doi: 10.1016/s0035-9203(02)90297-x. PMID 12055810
- [Background] MCGREGOR IA, GILLES HM, WALTERS JH, DAVIES AH, PEARSON FA. Effects of heavy and repeated malarial infections on Gambian infants and children; effects of erythrocytic parasitization. Br Med J. 1956 Sep 22;2(4994):686-92. doi: 10.1136/bmj.2.4994.686. No abstract available. PMID 13356045
- [Background] Meis JF, Ponnudurai T, Mons B, van Belkum A, van Eerd PM, Druilhe P, Schellekens H. Plasmodium falciparum: studies on mature exoerythrocytic forms in the liver of the chimpanzee, Pan troglodytes. Exp Parasitol. 1990 Jan;70(1):1-11. doi: 10.1016/0014-4894(90)90080-v. PMID 2403931
- [Background] Mendis K, Sina BJ, Marchesini P, Carter R. The neglected burden of Plasmodium vivax malaria. Am J Trop Med Hyg. 2001 Jan-Feb;64(1-2 Suppl):97-106. doi: 10.4269/ajtmh.2001.64.97. PMID 11425182
- [Background] Ministerio de Salud, Republica de Colombia. 2000. Guía de atención de la malariahttp://www.metrosalud.gov.co/Paginas/Protocolos/MinSalud/guias/31-MALARIA.htm.
- [Background] Ministerio de la Protección Social. República de Colombia. 2005. http://www.minproteccionsocial.gov.co/MseContent/images/news/DocNewsNo603701.pdf
- [Background] Nardin E, Clavijo P, Mons B, van Belkum A, Ponnudurai T, Nussenzweig RS. T cell epitopes of the circumsporozoite protein of Plasmodium vivax. Recognition by lymphocytes of a sporozoite-immunized chimpanzee. J Immunol. 1991 Mar 1;146(5):1674-8. PMID 1704402
- [Background] NCI.,NIH., DCTD., DHHS. Common Terminology Criteria for Adverse Events v3.0. 2003. http://ctep.cancer.gov/forms/CTCAEv3.pdf
- [Background] Nosten F, McGready R, Simpson JA, Thwai KL, Balkan S, Cho T, Hkirijaroen L, Looareesuwan S, White NJ. Effects of Plasmodium vivax malaria in pregnancy. Lancet. 1999 Aug 14;354(9178):546-9. doi: 10.1016/s0140-6736(98)09247-2. PMID 10470698
- [Background] OMS. 2005. World Malaria Report 2005. Prepared by Roll Back Malaria, WHO and Unicef. http://www.rbm.who.int/wmr2005/pdf/WMReport_lr.pdf.
- [Background] Padilla, JC., Guhl, F., Soto, J., Alvarez, G. Diagnóstico y terapéutica de las enfermedades transmitidas por vectores en Colombia.1999, v.2500. p.128
- [Background] Perlaza BL, Zapata C, Valencia AZ, Hurtado S, Quintero G, Sauzet JP, Brahimi K, Blanc C, Arevalo-Herrera M, Druilhe P, Herrera S. Immunogenicity and protective efficacy of Plasmodium falciparum liver-stage Ag-3 in Aotus lemurinus griseimembra monkeys. Eur J Immunol. 2003 May;33(5):1321-7. doi: 10.1002/eji.200323339. PMID 12731057
- [Background] Phillips-Howard PA. Epidemiological and control issues related to malaria in pregnancy. Ann Trop Med Parasitol. 1999 Dec;93 Suppl 1:S11-7. doi: 10.1080/00034989957691. PMID 10715684
- [Background] Powell RD, McNamara JV. Infection with chloroquine-resistant Plasmodium falciparum in man: prepatent periods, incubation periods, and relationships between parasitemia and the onset of fever in nonimmune persons. Ann N Y Acad Sci. 1970 Oct 30;174(2):1027-41. doi: 10.1111/j.1749-6632.1970.tb45625.x. No abstract available. PMID 4993529
- [Background] Rieckmann KH. Human immunization with attenuated sporozoites. Bull World Health Organ. 1990;68 Suppl(Suppl):13-6. PMID 2094578
- [Background] Rieckmann KH, Beaudoin RL, Cassells JS, Sell KW. Use of attenuated sporozoites in the immunization of human volunteers against falciparum malaria. Bull World Health Organ. 1979;57 Suppl 1(Suppl):261-5. PMID 120773
- [Background] Salas ML, Romero JF, Solarte Y, Olano V, Herrera MA, Herrera S. Development of sporogonic cycle of Plasmodium vivax in experimentally infected Anopheles albimanus mosquitoes. Mem Inst Oswaldo Cruz. 1994;89 Suppl 2:115-9. doi: 10.1590/s0074-02761994000600024. PMID 7565121
- [Background] Singh N, Shukla MM, Sharma VP. Epidemiology of malaria in pregnancy in central India. Bull World Health Organ. 1999;77(7):567-72. PMID 10444880
- [Background] Snounou G, Viriyakosol S, Jarra W, Thaithong S, Brown KN. Identification of the four human malaria parasite species in field samples by the polymerase chain reaction and detection of a high prevalence of mixed infections. Mol Biochem Parasitol. 1993 Apr;58(2):283-92. doi: 10.1016/0166-6851(93)90050-8. PMID 8479452
- [Background] Soto J, Toledo J, Gutierrez P, Luzz M, Llinas N, Cedeno N, Dunne M, Berman J. Plasmodium vivax clinically resistant to chloroquine in Colombia. Am J Trop Med Hyg. 2001 Aug;65(2):90-3. doi: 10.4269/ajtmh.2001.65.90. PMID 11508397
- [Background] Talisuna AO, Bloland P, D'Alessandro U. History, dynamics, and public health importance of malaria parasite resistance. Clin Microbiol Rev. 2004 Jan;17(1):235-54. doi: 10.1128/CMR.17.1.235-254.2004. PMID 14726463
- [Background] Trigg, PI., and Kondrachine, AV. 1998. The current global malaria situation, p. 11-22. In I. Sherman (ed.), Malaria: Parasite biology, pathogenesis and protection. AMS Press, Washington DC.
- [Background] Valderrama-Aguirre A, Quintero G, Gomez A, Castellanos A, Perez Y, Mendez F, Arevalo-Herrera M, Herrera S. Antigenicity, immunogenicity, and protective efficacy of Plasmodium vivax MSP1 PV200l: a potential malaria vaccine subunit. Am J Trop Med Hyg. 2005 Nov;73(5 Suppl):16-24. doi: 10.4269/ajtmh.2005.73.16. PMID 16291762
- [Background] Wilairatana P, Krudsood S, Treeprasertsuk S, Chalermrut K, Looareesuwan S. The future outlook of antimalarial drugs and recent work on the treatment of malaria. Arch Med Res. 2002 Jul-Aug;33(4):416-21. doi: 10.1016/s0188-4409(02)00371-5. PMID 12234533
- [Background] Walther M, Dunachie S, Keating S, Vuola JM, Berthoud T, Schmidt A, Maier C, Andrews L, Andersen RF, Gilbert S, Poulton I, Webster D, Dubovsky F, Tierney E, Sarpotdar P, Correa S, Huntcooke A, Butcher G, Williams J, Sinden RE, Thornton GB, Hill AV. Safety, immunogenicity and efficacy of a pre-erythrocytic malaria candidate vaccine, ICC-1132 formulated in Seppic ISA 720. Vaccine. 2005 Jan 4;23(7):857-64. doi: 10.1016/j.vaccine.2004.08.020. PMID 15603885
- [Background] Yagmur Y, Kara IH, Aldemir M, Buyukbayram H, Tacyildiz IH, Keles C. Spontaneous rupture of malarial spleen: two case reports and review of literature. Crit Care. 2000;4(5):309-13. doi: 10.1186/cc713. Epub 2000 Aug 10. PMID 11056757
- [Background] Zapata JC, Perlaza BL, Hurtado S, Quintero GE, Jurado D, Gonzalez I, Druilhe P, Arevalo-Herrera M, Herrera S. Reproducible infection of intact Aotus lemurinus griseimembra monkeys by Plasmodium falciparum sporozoite inoculation. J Parasitol. 2002 Aug;88(4):723-9. doi: 10.1645/0022-3395(2002)088[0723:RIOIAL]2.0.CO;2. PMID 12197121
- See also: Institutional Site — http://www.inmuno.org
- See also: register clinical trials — http://www.clinicaltrials.gov
- See also: World Health Organization — http://www.who.int/es

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 18
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 2 | 9
  Male | 1 | 4 | 4 | 9
Region of Enrollment [Number; unit: participants]
  Colombia | 6 | 6 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (11) | 23 (2) | 27 (5) | 27 (7)

OUTCOME MEASURES:

1. Primary Outcome: Infection for P. Vivax
Description: Thick blood smear was performed to patients daily on days 7 to 23, and every other day until day 29. Any prove of P. vivax infection was considered positive and confirmed later by real time polymerase chain reaction (rPCR).
Time Frame: Twenty eight days
Population: Values in the data table represent time to occurrence of P.Vivax infection (prepatent period).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 6 | 6 | 6
days | 11 (2) | 11 (1) | 9 (4)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Volunteers were directly observed by a study physician for one hour post-challenge, they were phone called approximately eight hours after challenge to control her/his evolution and then were followed by by the physician at day 1 after challenge.
Arm/Group | Group 1 | Group 2 | Group 3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 4/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=6) | Group 2 (N=6) | Group 3 (N=6)
Local pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 1 (1)
Local edema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Local erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Arm pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less